CLINICAL TRIAL: NCT01845818
Title: Observational Study in AS and PsA Patients to Evaluate Work Productivity Before and After the Start of Adalimumab Therapy in Daily Practice in Belgium
Brief Title: Study in Ankylosing Spondylitis (AS) and Psoriatic Arthritis (PsA) Patients to Evaluate Work Productivity Before and After the Start of Adalimumab Therapy in Daily Practice in Belgium
Acronym: SPACTIVE
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P13-990
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Results first posted 2019-01-09 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2018-05

CONDITIONS: Ankylosing Spondylitis; Psoriatic Arthritis
Keywords: work productivity; multicenter study
MeSH Terms: conditions — Spondylitis, Ankylosing; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ankylosing Spondylitis and Psoriatic Arthritis: Participants with AS and PsA and in whom adalimumab treatment is initiated. All medication will be prescribed in the usual manner in accordance with the terms of the marketing authorization and in line with the Belgian reimbursement criteria.

SUMMARY:
This observational study will document to what extent in daily clinical practice the work productivity is affected before and after the start of adalimumab treatment.

Changes in the employment status and work productivity of participants with AS and PsA before and after the start of adalimumab will be noted. The relationship between employment status, work productivity, disease activity and clinical evaluations will be evaluated. Since AS and PsA might be diseases with a strong impact on the daily life of the participant, an evaluation will be performed to the effect of the disease on quality of life and work productivity.

ELIGIBILITY:
Inclusion Criteria:

* Patient >= 18 years and <= 50 years
* Patient diagnosed with AS or PsA
* Patient to be initiated on adalimumab (according to the Marketing Authorization and Belgian reimbursement criteria)
* Patient willing to sign informed consent

Exclusion Criteria:

* Any contraindication for adalimumab as specified in the corresponding Summary of Product Characteristics (SmPC)
* Patient previously treated with biologics
* Patient participating in other AbbVie-sponsored trials

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants with AS and PsA followed in university or peripheral hospitals or peripheral private practices with experience in AS and PsA care.
Sampling Method: Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2013-06-05 (Actual); Primary Completion 2017-06-23 (Actual); Study Completion 2017-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Ankylosing Spondylitis: Participants with ankylosing spondylitis and in whom adalimumab treatment is initiated.
- Psoriatic Arthritis: Participants with psoriatic arthritis and in whom adalimumab treatment is initiated.
Period: Overall Study
Arm/Group | Ankylosing Spondylitis | Psoriatic Arthritis
Started | 126 | 57
Completed | 81 | 40
Not Completed | 45 | 17
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 7 | 5
Not completed — Administrative Reasons | 3 | 1
Not completed — Serious Adverse Event | 1 | 1
Not completed — Other | 25 | 8
Not completed — Did Not Receive Any Dose of Adalimumab | 5 | 0
Not completed — No Follow-Up Data Available | 4 | 1

BASELINE CHARACTERISTICS:
Population: Participants who not receive any dose of adalimumab and those who had no follow-up data available (see Participant Flow) are not included.
Groups:
- Ankylosing Spondylitis: Participants with ankylosing spondylitis and in whom adalimumab treatment was initiated.
- Psoriatic Arthritis: Participants with psoriatic arthritis and in whom adalimumab treatment was initiated.
- Total: Total of all reporting groups
Arm/Group | Ankylosing Spondylitis | Psoriatic Arthritis | Total
Number analyzed (Participants) | 117 | 56 | 173
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.74 (9.55) | 43.32 (8.39) | 39.54 (9.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 28 | 87
  Male | 58 | 28 | 86
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 114 | 55 | 169
  Other (Not Specified) | 2 | 0 | 2
  Missing | 1 | 1 | 2
Total Work Productivity Impairment (TWPI) [Mean (Standard Deviation); unit: percentage of TWPI] — Mean percentage of TWPI due to disease (based on the Work Productivity and Activity Impairment [WPAI] questionnaire) is presented, calculated as: Absenteeism (%) + extent to which disease decreased productivity (%)* [number of hours worked / (number of hours of work missed due to disease + number of hours worked)]. WPAI is a questionnaire used to evaluate lost productivity; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity. Population: Participants with a questionnaire completed at baseline are included.
  percentage of TWPI
    number analyzed (Participants) | 64 | 33 | 97
    (all) | 57.09 (27.47) | 47.54 (31.86) | 53.84 (29.23)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Month 18 in TWPI Due to Disease (Ankylosing Spondylitis and Psoriatic Arthritis Combined)
Description: The mean percentage of TWPI due to disease (based on the WPAI questionnaire) is presented, calculated as: Absenteeism (%) + extent to which disease decreased productivity (%)* [number of hours worked / (number of hours of work missed due to disease + number of hours worked)]. WPAI is a questionnaire used to evaluate lost productivity; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity. "Change" was calculated as the value at baseline minus the value at Month 18.
Time Frame: Baseline, Month 18
Population: Per Protocol Set: all participants enrolled in the study who received at least one dose of adalimumab, who had no major protocol deviations, and for whom any follow-up data were available. Participants with professional activity and with a questionnaire completed at given time point are included.
Measure: Mean (Standard Deviation); unit: percentage of TWPI
Groups:
- Ankylosing Spondylitis and Psoriatic Arthritis: Participants with ankylosing spondylitis and psoriatic arthritis in whom adalimumab treatment was initiated.
Arm/Group | Ankylosing Spondylitis and Psoriatic Arthritis
Number analyzed (Participants) | 56
percentage of TWPI | -29.15 (35.37)

2. Secondary Outcome: Change From Baseline at Month 18 in TWPI Due to Disease (Ankylosing Spondylitis and Psoriatic Arthritis Separately)
Description: as for outcome 1
Time Frame: Baseline, Month 18
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of TWPI
Groups:
- Ankylosing Spondylitis: Participants with ankylosing spondylitis in whom adalimumab treatment was initiated.
- Psoriatic Arthritis: Participants with psoriatic arthritis in whom adalimumab treatment was initiated.
Arm/Group | Ankylosing Spondylitis | Psoriatic Arthritis
Number analyzed (Participants) | 39 | 17
percentage of TWPI | -30.47 (34.88) | -26.11 (37.39)

3. Secondary Outcome: Number of Participants Employed at Each Assessed Visit
Description: As assessed by the WPAI questionnaire, a questionnaire used to evaluate lost work productivity due to disease (yes=employed; no=not employed). Last observation is the last observation after baseline at which any of the questionnaire items was completed.
Time Frame: Baseline, Months 3, 6, 12, 18
Population: Per Protocol Set: all participants enrolled in the study who received at least one dose of adalimumab, who had no major protocol deviations, and for whom any follow-up data were available. Participants with a questionnaire completed at given time point are included.
Measure: Count of Participants; unit: Participants
Groups:
- Ankylosing Spondylitis and Psoriatic Arthritis: Participants with ankylosing spondylitis or psoriatic arthritis in whom adalimumab treatment was initiated.
Arm/Group | Ankylosing Spondylitis | Psoriatic Arthritis | Ankylosing Spondylitis and Psoriatic Arthritis
Number analyzed (Participants) | 112 | 55 | 167
Participants
  Baseline : No | 26 | 14 | 40
  Baseline : Yes | 86 | 41 | 127
  Baseline : All | 112 | 55 | 167
  Month 3 : No: number analyzed (Participants) | 99 | 48 | 147
  Month 3 : No | 21 | 10 | 31
  Month 3 : Yes: number analyzed (Participants) | 99 | 48 | 147
  Month 3 : Yes | 78 | 38 | 116
  Month 3 : All: number analyzed (Participants) | 99 | 48 | 147
  Month 3 : All | 99 | 48 | 147
  Month 6 : No: number analyzed (Participants) | 87 | 44 | 131
  Month 6 : No | 17 | 10 | 27
  Month 6 : Yes: number analyzed (Participants) | 87 | 44 | 131
  Month 6 : Yes | 70 | 34 | 104
  Month 6 : All: number analyzed (Participants) | 87 | 44 | 131
  Month 6 : All | 87 | 44 | 131
  Month 12 : No: number analyzed (Participants) | 81 | 38 | 119
  Month 12 : No | 14 | 8 | 22
  Month 12 : Yes: number analyzed (Participants) | 81 | 38 | 119
  Month 12 : Yes | 67 | 30 | 97
  Month 12 : All: number analyzed (Participants) | 81 | 38 | 119
  Month 12 : All | 81 | 38 | 119
  Month 18 : No: number analyzed (Participants) | 71 | 39 | 110
  Month 18 : No | 12 | 8 | 20
  Month 18 : Yes: number analyzed (Participants) | 71 | 39 | 110
  Month 18 : Yes | 59 | 31 | 90
  Month 18 : All: number analyzed (Participants) | 71 | 39 | 110
  Month 18 : All | 71 | 39 | 110
  Last Observation : No: number analyzed (Participants) | 108 | 55 | 163
  Last Observation : No | 21 | 13 | 34
  Last Observation : Yes: number analyzed (Participants) | 108 | 55 | 163
  Last Observation : Yes | 87 | 42 | 129
  Last Observation : All: number analyzed (Participants) | 108 | 55 | 163
  Last Observation : All | 108 | 55 | 163

4. Secondary Outcome: Percentage of Missed Working Hours (Absenteeism) Due to Disease 7 Days Prior to Each Visit
Description: Absenteeism, presented as the mean percentage of work time missed due to disease (as reported on the WPAI), and calculated as: 100*number of hours of work missed due to disease / (number of hours of work missed due to disease + number of hours worked). WPAI is a questionnaire used to evaluate lost productivity; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity. Last observation is the last observation after baseline at which any of the questionnaire items was completed.
Time Frame: Baseline, Months 3, 6, 12, 18
Population: Per Protocol Set: all participants enrolled in the study who received at least one dose of adalimumab, who had no major protocol deviations, and for whom any follow-up data were available. Participants with a professional activity and with a questionnaire completed at given time point are included.
Measure: Mean (Standard Deviation); unit: percentage of work time missed
Arm/Group | Ankylosing Spondylitis | Psoriatic Arthritis | Ankylosing Spondylitis and Psoriatic Arthritis
Number analyzed (Participants) | 76 | 35 | 110
percentage of work time missed
  Baseline: number analyzed (Participants) | 73 | 35 | 108
  Baseline | 24.29 (40.09) | 12.27 (27.76) | 20.39 (36.86)
  Month 3: number analyzed (Participants) | 65 | 34 | 99
  Month 3 | 10.24 (29.53) | 5.39 (19.56) | 8.57 (26.53)
  Month 6: number analyzed (Participants) | 62 | 33 | 95
  Month 6 | 6.79 (21.45) | 5.82 (19.58) | 6.45 (20.72)
  Month 12: number analyzed (Participants) | 61 | 22 | 83
  Month 12 | 5.90 (21.00) | 2.27 (10.66) | 4.94 (18.83)
  Month 18: number analyzed (Participants) | 54 | 25 | 79
  Month 18 | 12.19 (31.34) | 2.00 (10.00) | 8.97 (26.85)
  Last Observation: number analyzed (Participants) | 76 | 34 | 110
  Last Observation | 12.94 (31.71) | 4.41 (18.94) | 10.31 (28.57)

5. Secondary Outcome: Percentage of Activity Impairment Due to Disease During the 7 Days Prior to Each Visit
Description: Activity impairment due to disease (the extent to which disease affected the ability to perform usual daily activities, as reported on the WPAI) is presented as the mean percentage of activity impairment, calculated as 100*scale value of WPAI question 6 (between 0 and 10) / 10. WPAI is a questionnaire used to evaluate lost productivity; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity. Last observation is the last observation after baseline at which any of the questionnaire items was completed.
Time Frame: Baseline, Months 3, 6, 12, 18
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage activity impairment
Arm/Group | Ankylosing Spondylitis | Psoriatic Arthritis | Ankylosing Spondylitis and Psoriatic Arthritis
Number analyzed (Participants) | 111 | 55 | 163
percentage activity impairment
  Baseline: number analyzed (Participants) | 111 | 51 | 162
  Baseline | 62.25 (22.75) | 57.25 (26.01) | 60.68 (23.86)
  Month 3: number analyzed (Participants) | 98 | 45 | 143
  Month 3 | 39.59 (28.68) | 32.22 (27.21) | 37.27 (28.34)
  Month 6: number analyzed (Participants) | 87 | 43 | 130
  Month 6 | 31.61 (26.05) | 33.72 (27.95) | 32.31 (26.60)
  Month 12: number analyzed (Participants) | 83 | 38 | 121
  Month 12 | 31.33 (26.22) | 30.00 (29.50) | 30.91 (27.17)
  Month 18: number analyzed (Participants) | 71 | 39 | 110
  Month 18 | 28.59 (27.89) | 25.13 (28.46) | 27.36 (28.01)
  Last Observation: number analyzed (Participants) | 108 | 55 | 163
  Last Observation | 34.17 (28.75) | 32.73 (29.22) | 33.68 (28.82)

6. Secondary Outcome: Percentage of Impairment While Working Due to Disease (Presenteeism) 7 Days Prior to Each Visit
Description: As measured by the WPAI-Specific Health Problem questionnaire. Presenteeism (the extent to which disease decreased productivity, as reported on the WPAI) is presented as the mean percentage of impairment while working due to disease, and calculated as: 100*scale value of question 5 on the WPAI (between 0 and 10) / 10. WPAI is a questionnaire used to evaluate lost productivity; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity. Last observation is the last observation after baseline at which any of the questionnaire items was completed.
Time Frame: Baseline, Months 3, 6, 12, 18
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage impairment while working
Arm/Group | Ankylosing Spondylitis | Psoriatic Arthritis | Ankylosing Spondylitis and Psoriatic Arthritis
Number analyzed (Participants) | 75 | 36 | 111
percentage impairment while working
  Baseline: number analyzed (Participants) | 66 | 34 | 100
  Baseline | 55.45 (25.91) | 46.18 (30.35) | 52.30 (27.70)
  Month 3: number analyzed (Participants) | 63 | 34 | 97
  Month 3 | 24.44 (24.48) | 26.18 (27.53) | 25.05 (25.46)
  Month 6: number analyzed (Participants) | 60 | 32 | 92
  Month 6 | 22.67 (19.30) | 28.75 (29.04) | 24.78 (23.18)
  Month 12: number analyzed (Participants) | 60 | 23 | 83
  Month 12 | 25.17 (24.11) | 15.65 (20.41) | 22.53 (23.42)
  Month 18: number analyzed (Participants) | 52 | 28 | 80
  Month 18 | 25.00 (27.97) | 19.29 (25.81) | 23.00 (27.21)
  Last Observation | 28.93 (29.25) | 26.39 (28.40) | 28.11 (28.87)

7. Secondary Outcome: Health Assessment Questionnaire-Disability Index (HAQ-DI) Scores Over Time (Psoriatic Arthritis)
Description: The HAQ-DI is a self-reported assessment of how the participant's disease affects their ability to function in their daily life over the past week. The HAQ-DI for a participant is calculated as the mean of the following 8 category scores: dressing and grooming, rising, eating, walking, hygiene, reach, grip, and activities. Scores range from 0 to 3, with a lower score demonstrating less disability. Last observation is the last observation after baseline at which any of the questionnaire items was completed.
Time Frame: Baseline, Months 3, 6, 12, 18
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 55
units on a scale
  Baseline | 1.34 (0.58)
  Month 3: number analyzed (Participants) | 47
  Month 3 | 0.70 (0.57)
  Month 6: number analyzed (Participants) | 45
  Month 6 | 0.70 (0.61)
  Month 12: number analyzed (Participants) | 41
  Month 12 | 0.62 (0.65)
  Month 18: number analyzed (Participants) | 41
  Month 18 | 0.54 (0.57)
  Last Observation: number analyzed (Participants) | 54
  Last Observation | 0.68 (0.61)

8. Secondary Outcome: Dermatology Life Quality Index (DLQI) Scores Over Time (Psoriatic Arthritis)
Description: The DLQI score is a participant-reported outcome consisting of a set of 10 questions regarding the degree to which the participant's skin has affected certain behaviors and quality of life over the last week. Responses to each are: very much (score of 3), a lot, a little, or not at all (score of 0); responses are summed. The DLQI score ranges from 0 (best) to 30 (worst); the higher the score, the more quality of life is impaired. Last observation is the last observation after baseline at which any of the questionnaire items was completed.
Time Frame: Baseline, Months 3, 6, 12, 18
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 55
units on a scale
  Baseline | 5.85 (7.25)
  Month 3: number analyzed (Participants) | 47
  Month 3 | 3.11 (5.72)
  Month 6: number analyzed (Participants) | 42
  Month 6 | 3.29 (6.93)
  Month 12: number analyzed (Participants) | 37
  Month 12 | 2.30 (4.81)
  Month 18: number analyzed (Participants) | 40
  Month 18 | 2.08 (4.84)
  Last Observation: number analyzed (Participants) | 54
  Last Observation | 3.24 (6.40)

9. Secondary Outcome: Health Assessment Questionnaire Modified for Spondyloarthropathies (HAQ-S) Scores Over Time (Ankylosing Spondylitis)
Description: The HAQ-S is a self-reported measure to assess the physical function and health-related quality of life. The Disability Index (DI) of HAQ-S is calculated as the mean of the following 8 category scores (range: 0 [without any difficulty] to 3 [unable to do]): Dressing and Grooming, Rising, Eating, Walking, Hygiene, Reach, Grip, and Activities. Five additional items in the functional status measure were included in the HAQ-S, including carrying heavy packages, sitting for long periods, able to work at a flat topped table, and (if the participant had a driver's license or a car) able to look in the rear view mirror and able to turn head to drive in reverse. The overall score ranges from 0 (no disability) to 3 (very severe, high-dependency disability). Last observation is the last observation after baseline at which any of the questionnaire items was completed.
Time Frame: Baseline, Months 3, 6, 12, 18
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 114
units on a scale
  Baseline | 1.21 (0.48)
  Month 3: number analyzed (Participants) | 96
  Month 3 | 0.76 (0.50)
  Month 6: number analyzed (Participants) | 88
  Month 6 | 0.59 (0.48)
  Month 12: number analyzed (Participants) | 86
  Month 12 | 0.60 (0.48)
  Month 18: number analyzed (Participants) | 70
  Month 18 | 0.61 (0.53)
  Last Observation: number analyzed (Participants) | 105
  Last Observation | 0.68 (0.54)

10. Secondary Outcome: Disease Activity Score 28 (DAS-28) Over Time (Psoriatic Arthritis)
Description: The DAS-28 is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, erythrocyte sedimentation rate (ESR), and the Subject's Global Assessment of Disease Activity (subject rates disease activity using a Likert scale from 0 [low activity] to 10 [high activity]) are included in the DAS-28 score. Scores on the DAS-28 range from 0 to 10. A DAS-28 score > 5.1 indicates high disease activity, a DAS-28 score < 3.2 indicates low disease activity, and a DAS-28 score < 2.6 indicates clinical remission. Last observation is the last observation after baseline at which any of the questionnaire items was completed.
Time Frame: Baseline, Months 3, 6, 12, 18
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 33
units on a scale
  Baseline: number analyzed (Participants) | 30
  Baseline | 4.37 (1.03)
  Month 3: number analyzed (Participants) | 22
  Month 3 | 2.26 (1.04)
  Month 6: number analyzed (Participants) | 17
  Month 6 | 2.17 (1.19)
  Month 12: number analyzed (Participants) | 18
  Month 12 | 1.99 (1.06)
  Month 18: number analyzed (Participants) | 17
  Month 18 | 1.99 (1.01)
  Last Observation | 2.05 (1.19)

11. Secondary Outcome: Percentage of Body Surface Area (BSA) Affected Over Time (Psoriatic Arthritis)
Description: Percentage of BSA affected by psoriatic arthritis was assessed by clinical evaluation. Last observation is the last observation after baseline at which any of the questionnaire items was completed.
Time Frame: Baseline, Months 3, 6, 12, 18
Population: Per Protocol Set: all participants enrolled in the study who received at least one dose of adalimumab, who had no major protocol deviations, and for whom any follow-up data were available. Participants with a BSA assessment at given time point are included.
Measure: Number; unit: percentage of participants
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 56
percentage of participants
  Baseline: 0%: number analyzed (Participants) | 55
  Baseline: 0% | 34.5
  Baseline: < 3%: number analyzed (Participants) | 55
  Baseline: < 3% | 32.7
  Baseline: 3% to 10%: number analyzed (Participants) | 55
  Baseline: 3% to 10% | 27.3
  Baseline: 11% to 20%: number analyzed (Participants) | 55
  Baseline: 11% to 20% | 5.5
  Baseline: > 20%: number analyzed (Participants) | 55
  Baseline: > 20% | 0.0
  Month 3: 0%: number analyzed (Participants) | 50
  Month 3: 0% | 52.0
  Month 3: < 3%: number analyzed (Participants) | 50
  Month 3: < 3% | 36.0
  Month 3: 3% to 10%: number analyzed (Participants) | 50
  Month 3: 3% to 10% | 8.0
  Month 3: 11% to 20%: number analyzed (Participants) | 50
  Month 3: 11% to 20% | 2.0
  Month 3: > 20%: number analyzed (Participants) | 50
  Month 3: > 20% | 2.0
  Month 6: 0%: number analyzed (Participants) | 50
  Month 6: 0% | 56.0
  Month 6: < 3%: number analyzed (Participants) | 50
  Month 6: < 3% | 36.0
  Month 6: 3% to 10%: number analyzed (Participants) | 50
  Month 6: 3% to 10% | 8.0
  Month 6: 11% to 20%: number analyzed (Participants) | 50
  Month 6: 11% to 20% | 0.0
  Month 6: > 20%: number analyzed (Participants) | 50
  Month 6: > 20% | 0.0
  Month 12: 0%: number analyzed (Participants) | 44
  Month 12: 0% | 59.1
  Month 12: < 3%: number analyzed (Participants) | 44
  Month 12: < 3% | 36.4
  Month 12: 3% to 10%: number analyzed (Participants) | 44
  Month 12: 3% to 10% | 4.5
  Month 12: 11% to 20%: number analyzed (Participants) | 44
  Month 12: 11% to 20% | 0.0
  Month 12: > 20%: number analyzed (Participants) | 44
  Month 12: > 20% | 0.0
  Month 18: 0%: number analyzed (Participants) | 41
  Month 18: 0% | 63.4
  Month 18: < 3%: number analyzed (Participants) | 41
  Month 18: < 3% | 31.7
  Month 18: 3% to 10%: number analyzed (Participants) | 41
  Month 18: 3% to 10% | 2.4
  Month 18: 11% to 20%: number analyzed (Participants) | 41
  Month 18: 11% to 20% | 2.4
  Month 18: > 20%: number analyzed (Participants) | 41
  Month 18: > 20% | 0.0
  Last Observation: 0% | 60.7
  Last Observation: < 3% | 30.4
  Last Observation: 3% to 10% | 5.4
  Last Observation: 11% to 20% | 1.8
  Last Observation: > 20% | 1.8

12. Secondary Outcome: Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Scores Over Time (Ankylosing Spondylitis)
Description: The BASDAI is used for measuring and evaluating disease activity in ankylosing spondylitis. This index consists of 6 questions pertaining to the 5 major symptoms of ankylosing spondylitis: fatigue, spinal pain, joint pain/swelling, areas of localized tenderness (or enthesitis, defined as inflammation of tendons and ligaments), duration of morning stiffness, severity of morning stiffness. A visual analogue scale ranging from 0 (none) to 10 (very severe) is used to answer the questions. The final BASDAI score averages the individual assessments for a final score range of 0 to 10 (0 being no problem and 10 being the worst problem). Last observation is the last observation after baseline at which any of the questionnaire items was completed.
Time Frame: Baseline, Months 3, 6, 12, 18
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 116
units on a scale
  Baseline | 6.85 (1.32)
  Month 3: number analyzed (Participants) | 103
  Month 3 | 3.97 (2.27)
  Month 6: number analyzed (Participants) | 90
  Month 6 | 3.18 (2.01)
  Month 12: number analyzed (Participants) | 88
  Month 12 | 3.27 (2.37)
  Month 18: number analyzed (Participants) | 73
  Month 18 | 3.09 (2.21)
  Last Observation: number analyzed (Participants) | 110
  Last Observation | 3.76 (2.50)

13. Secondary Outcome: Acute Phase Reactant: Erythrocyte Sedimentation Rate (ESR) Values Over Time
Description: The ESR is a practicable and sensitive but not specific parameter for measuring disease progression. By means of the ESR it can be generally distinguished between an active and nonactive rheumatic disease. The normal reference range is, as a rule, 0 to 10 mm/h for men and 0 to 15 mm/h for women. The higher the ESR value out of the normal range, the higher is the disease activity. Last observation is the last observation after baseline at which an assessment was completed.
Time Frame: Baseline, Months 3, 6, 12, 18
Population: Per Protocol Set: all participants enrolled in the study who received at least one dose of adalimumab, who had no major protocol deviations, and for whom any follow-up data were available. Participants with an assessment at given time point are included.
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | Ankylosing Spondylitis | Psoriatic Arthritis | Ankylosing Spondylitis and Psoriatic Arthritis
Number analyzed (Participants) | 80 | 47 | 126
mm/h
  Baseline: number analyzed (Participants) | 79 | 47 | 126
  Baseline | 15.14 (14.74) | 12.77 (12.05) | 14.25 (13.80)
  Month 3: number analyzed (Participants) | 66 | 40 | 106
  Month 3 | 8.23 (8.13) | 6.05 (5.17) | 7.41 (7.21)
  Month 6: number analyzed (Participants) | 65 | 36 | 101
  Month 6 | 7.65 (7.15) | 10.83 (13.62) | 8.78 (10.00)
  Month 12: number analyzed (Participants) | 52 | 36 | 88
  Month 12 | 7.38 (8.54) | 10.03 (11.86) | 8.47 (10.05)
  Month 18: number analyzed (Participants) | 49 | 29 | 78
  Month 18 | 7.63 (6.84) | 7.17 (5.98) | 7.46 (6.50)
  Last Observation: number analyzed (Participants) | 80 | 45 | 125
  Last Observation | 8.19 (6.93) | 10.84 (12.49) | 9.14 (9.36)

14. Secondary Outcome: Acute Phase Reactant: C-Reactive Protein (CRP) Values Over Time
Description: CRP is an acute phase reactant plasma protein, normally produced by the liver, which is commonly used as an indirect measure of the extent and activity of an inflammation. The CRP normal reference range in the blood is, as a rule, from 0 to 1.0 mg/dL. Last observation is the last observation after baseline at which an assessment was completed.
Time Frame: Baseline, Months 3, 6, 12, 18
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ankylosing Spondylitis | Psoriatic Arthritis | Ankylosing Spondylitis and Psoriatic Arthritis
Number analyzed (Participants) | 108 | 51 | 159
mg/dL
  Baseline | 2.36 (7.16) | 1.48 (3.06) | 2.08 (6.15)
  Month 3: number analyzed (Participants) | 76 | 42 | 118
  Month 3 | 0.35 (0.45) | 0.81 (1.95) | 0.51 (1.23)
  Month 6: number analyzed (Participants) | 74 | 38 | 112
  Month 6 | 0.62 (1.18) | 0.82 (2.08) | 0.69 (1.54)
  Month 12: number analyzed (Participants) | 63 | 40 | 103
  Month 12 | 0.39 (0.50) | 0.66 (1.66) | 0.49 (1.11)
  Month 18: number analyzed (Participants) | 60 | 33 | 93
  Month 18 | 0.50 (0.76) | 0.36 (0.55) | 0.45 (0.69)
  Last Observation: number analyzed (Participants) | 100 | 50 | 150
  Last Observation | 0.52 (0.90) | 0.91 (2.04) | 0.65 (1.39)

15. Secondary Outcome: Physician's Assessment of Disease Activity Visual Analogue Scale (VAS) Scores Over Time
Description: The VAS score assessed by physicians was used to determine the disease activity of ankylosing spondylitis and psoriatic arthritis in the past week. The level of disease activity was measured in millimeters (mm) on a 100 mm horizontal line. The score ranged from 0 (none) to 100 (most disease activity).
Time Frame: Baseline, Months 3, 6, 12, 18
Population: Per Protocol Set: all participants enrolled in the study who received at least one dose of adalimumab, who had no major protocol deviations, and for whom any follow-up data were available. Participants with an assessment completed at given time point are included.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ankylosing Spondylitis | Psoriatic Arthritis | Ankylosing Spondylitis and Psoriatic Arthritis
Number analyzed (Participants) | 107 | 55 | 162
mm
  Baseline: number analyzed (Participants) | 106 | 52 | 158
  Baseline | 67.14 (16.03) | 59.35 (15.65) | 64.58 (16.28)
  Month 3: number analyzed (Participants) | 97 | 52 | 149
  Month 3 | 24.92 (20.51) | 21.19 (17.23) | 23.62 (19.45)
  Month 6: number analyzed (Participants) | 90 | 48 | 138
  Month 6 | 18.40 (17.57) | 19.34 (16.08) | 18.73 (17.01)
  Month 12: number analyzed (Participants) | 85 | 43 | 128
  Month 12 | 18.13 (17.76) | 17.12 (15.54) | 17.79 (17.00)
  Month 18: number analyzed (Participants) | 77 | 42 | 119
  Month 18 | 17.39 (18.03) | 15.07 (17.91) | 16.57 (17.95)
  Last Observation | 21.70 (21.00) | 18.31 (18.36) | 20.55 (20.15)

16. Secondary Outcome: Participant's Assessment of Disease Activity Visual Analogue Scale (VAS) Scores Over Time
Description: The VAS score assessed by participants was used to determine the disease activity of ankylosing spondylitis and psoriatic arthritis in the past week. The level of disease activity was measured in millimeters (mm) on a 100 mm horizontal line. The score ranged from 0 (none) to 100 (most disease activity).
Time Frame: Baseline, Months 3, 6, 12, 18
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ankylosing Spondylitis | Psoriatic Arthritis | Ankylosing Spondylitis and Psoriatic Arthritis
Number analyzed (Participants) | 113 | 55 | 168
mm
  Baseline | 67.53 (20.14) | 60.89 (19.91) | 65.36 (20.25)
  Month 3: number analyzed (Participants) | 100 | 50 | 150
  Month 3 | 36.31 (26.97) | 30.42 (25.58) | 34.35 (26.58)
  Month 6: number analyzed (Participants) | 90 | 46 | 136
  Month 6 | 25.80 (23.58) | 34.46 (28.63) | 28.73 (25.63)
  Month 12: number analyzed (Participants) | 85 | 39 | 124
  Month 12 | 28.89 (26.48) | 29.00 (27.39) | 28.93 (26.66)
  Month 18: number analyzed (Participants) | 71 | 40 | 111
  Month 18 | 24.86 (24.30) | 24.55 (25.30) | 24.75 (24.55)
  Last Observation: number analyzed (Participants) | 108 | 55 | 163
  Last Observation | 31.31 (26.95) | 32.64 (28.18) | 31.75 (27.29)

17. Secondary Outcome: Participant's Global Assessment of Pain VAS Scores Over Time
Description: The VAS score assessed by participants was used to determine the pain due to ankylosing spondylitis and psoriatic arthritis in the past week. The level of pain was measured in millimeters (mm) on a 100 mm horizontal line. The score ranged from 0 (no pain) to 100 (severe pain).
Time Frame: Baseline, Months 3, 6, 12, 18
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ankylosing Spondylitis | Psoriatic Arthritis | Ankylosing Spondylitis and Psoriatic Arthritis
Number analyzed (Participants) | 113 | 55 | 168
mm
  Baseline | 70.17 (18.59) | 64.24 (19.02) | 68.23 (18.88)
  Month 3: number analyzed (Participants) | 100 | 50 | 150
  Month 3 | 37.91 (27.63) | 29.60 (25.97) | 35.14 (27.28)
  Month 6: number analyzed (Participants) | 90 | 46 | 136
  Month 6 | 27.73 (24.49) | 34.93 (30.51) | 30.17 (26.78)
  Month 12: number analyzed (Participants) | 85 | 39 | 124
  Month 12 | 29.55 (26.80) | 30.79 (29.73) | 29.94 (27.64)
  Month 18: number analyzed (Participants) | 71 | 40 | 111
  Month 18 | 27.41 (25.84) | 25.68 (27.69) | 26.78 (26.41)
  Last Observation: number analyzed (Participants) | 108 | 55 | 163
  Last Observation | 33.35 (27.92) | 33.93 (30.69) | 33.55 (28.79)

ADVERSE EVENTS:
Time Frame: Up to 23 months plus 70 days. The average adalimumab treatment duration was 14.9 months (standard deviation: 5.6).
Description: Adverse events were analyzed for all participants as one group, per protocol.
Arm/Group | Ankylosing Spondylitis and Psoriatic Arthritis
All-Cause Mortality (participants affected / at risk) | 0/173
Serious Adverse Events (participants affected / at risk) | 1/173
Other Adverse Events (participants affected / at risk) | 0/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ankylosing Spondylitis and Psoriatic Arthritis (N=173)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2012-12-06): https://cdn.clinicaltrials.gov/large-docs/18/NCT01845818/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-04): https://cdn.clinicaltrials.gov/large-docs/18/NCT01845818/SAP_001.pdf